CLINICAL TRIAL: NCT07002970
Title: Combined Effect of Aerobic Exercise and Mediterranean Diet on Inflammatory Markers and Quality of Life in Obese Patients
Brief Title: Effect of Aerobic Exercise and Mediterranean Diet on Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Salah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P.T.REC/012/004630
Record Dates: First submitted 2025-05-23; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: aerobic exercise; inflammatory markers
MeSH Terms: conditions — Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): aerobic exercise program and Mediterranean diet
  Interventions: Other: aerobic exercise program; Other: Mediterranean diet
- control group (Active Comparator): Mediterranean diet
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: aerobic exercise program — All study group patients performed aerobic exercise on a treadmill. approved by the American College of Sports Medicine.
  Arms: study group
Other: Mediterranean diet — received a Mediterranean diet for 12 weeks tailored according to patients caloric needs

SUMMARY:
All study group patients performed aerobic exercise on a treadmill. approved by the American College of Sports Medicine.

Both groups received a Mediterranean diet for 12 weeks tailored according to patients' caloric needs

DETAILED DESCRIPTION:
All study group patients performed aerobic exercise on a treadmill approved by the American College of Sports Medicine. The program started with a warming-up phase through walking on a treadmill for 3-5 minutes at a slow speed. Then, 10-30 minutes of aerobic exercise training with moderate intensity (60-70% of maximum heart rate) and 10 minutes of cooling down with low speed and without inclination. Participants had 3 sessions/week for 3 months with close supervision of a physical therapist.

Both groups received a Mediterranean diet for 12 weeks tailored to patients' caloric needs. They received instructions about the consumption of olive oil as added lipid, the consumption of nuts and olives as snacks, daily high consumption of vegetables, fruits, and whole grains, dairy products, bi-weekly consumption of legumes, bi-weekly consumption of fish, and monthly consumption of meat. The main beneficial components of the Mediterranean diet are monounsaturated fats such as oleic acid in olive oil, polyunsaturated fats such as omega-3, high amounts of flavonoids and antioxidants found in fruits and vegetables, and high amounts of fiber found mainly in foods with a low glycemic index

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with BMI ranged from 30-39.9 kg/m 2.
* Their age was from 35 to 45 years old.
* Both genders.
* Stable vital signs (blood pressure, respiratory rate and temperature)
* Abdominal obesity measurements according to American heart association)
* Obese patients have one or more abnormal value of lipids profile.
* All patients with sedentary life style.
* All patients had insulin resistance

Exclusion Criteria:

* Rheumatic, neurologic, cardiovascular, respiratory, renal, lung problems, malignant tumors, and undiagnosed fever, which would prevent them from participating in aerobic exercises.
* Knee injury or knee surgery during the past six month or having a history of joint replacement or fracture or hereditary or acquired musculoskeletal disorders in lower limb.
* Major vision disorders.
* Drugs that would affect metabolism or balance.
* Assistive devices for walking.
* Pregnancy or breast feeding, and post-partum 12 months.
* Abdominal or rectal anus surgery.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Short Form Quality of Life Questionnaire (SF-36) | 12 weeks
  To measure the health related quality of life (HRQOL)in obese patient. SF-36 (version 2.0) is a 36-item measure of generic HRQOL in which 35 questions are transformed into eight dimensions; physical functioning, role limitation to physical problems, bodily pain, general health, vitality, social functioning, role limitations to emotional problems, and mental health Scores on all eight dimensions range from zero to 100, where higher scores represent better HRQOL

SECONDARY OUTCOMES:
Laboratory Measurements | 12 weeks
  After a 12-hour overnight fast, venous blood samples were collected from each participant in all participants before and after 12 weeks of treatment to measure, LDL, HDL, total cholesterol, TG levels milligrams per deciliter (mg/dL) and fasting blood glucose (FBG) measured in mg/dL (milligrams per deciliter) ,C-reactive protein (CRP) measured in milligrams per liter (mg/L), and (ESR) was measured in millimeters per hour (mm/hr) and fasting serum insulin measured and reported in micro International Units per milliliter (uIU/mL) by commercially available kits. All samples were drawn between 8 and 10 a.m. for later analysis.
Blood Pressure Measures | 12 weeks
  Systolic and diastolic blood pressures were measured for each participant before and after 12 weeks of treatment
body weight | 12 weeks
  Body weight was measured for each participant in kilograms
height | 12 weeks
  body height was measured for each participant in meters
waist and hip circumferences | 12 weeks
  waist and hip circumferences were measured for each participant in centimeter

CONTACTS AND LOCATIONS:
Overall Officials: mai salah, master, Principal Investigator — faculty of physical Cairo university
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt